CLINICAL TRIAL: NCT00055939
Title: A Phase II Study Of Intravenous DX-8951f (EXATECAN MESYLATE) Administered Daily For Five Days Every Three Weeks To Pediatric Patients With Relapsed Or Refractory Rhabdomyosarcoma
Brief Title: Exatecan Mesylate in Treating Children With Relapsed or Refractory Rhabdomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271888; DAIICHI-8951A-PRT033; SJCRH-DXRMS
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Sarcoma
Keywords: previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of exatecan mesylate in treating children who have relapsed or refractory rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate (complete and partial responses) in pediatric patients with relapsed or refractory rhabdomyosarcoma treated with exatecan mesylate.
* Determine the time to tumor progression in patients treated with this drug.
* Determine the median survival and survival at 6 and 12 months in patients treated with this drug.
* Assess pain in patients treated with this drug.
* Evaluate the quantitative and qualitative toxic effects of this drug in these patients.
* Evaluate the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive exatecan mesylate IV over 30 minutes on days 1-5. Treatment repeats every 3 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 6 additional courses beyond CR.

PROJECTED ACCRUAL: A total of 13-27 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or resistant rhabdomyosarcoma
* Measurable disease

  * The following are not considered measurable disease:

    * Ascites
    * Pleural effusion
    * Lytic bone lesions
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2 (over 10 years old)
* Lansky 60-100% (10 years old and under)

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 8.5 g/dL

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* Albumin at least 2.8 g/dL
* AST or ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)

Renal

* Creatinine no greater than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No life threatening illness (unrelated to tumor) within the past 6 months
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No concurrent active serious infection
* No concurrent uncontrolled infection
* No overt psychosis or other incompetency that would preclude study compliance or giving informed consent
* No other concurrent noncancer-related illness that would preclude study participation or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior autologous bone marrow or stem cell transplantation
* No concurrent anticancer biologic therapy

Chemotherapy

* Recovered from prior adjuvant or systemic chemotherapy
* Prior topoisomerase I inhibitor therapy allowed
* No other concurrent anticancer chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior extensive radiotherapy to the cranial-spinal axis, whole pelvis, or 25% of marrow reserve
* No concurrent anticancer radiotherapy

Surgery

* At least 4 weeks since prior major surgery
* Recovered from prior surgery
* No concurrent anticancer surgery

Other

* At least 28 days since prior investigational drugs (including analgesics or antiemetics)
* No more than 2 prior regimens for rhabdomyosarcoma
* No concurrent grapefruit-containing beverages or foods
* No other concurrent investigational drugs during and for 28 days after final dose of study drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (9):
- United States (8):
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada